CLINICAL TRIAL: NCT01467908
Title: Navigated Brain Stimulation in Diagnosis of Minimally Conscious State
Acronym: C-fMRI-NBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Institute of the Brain, Russia (Other)
Collaborators: City Hospital No 41, Ekaterinburg, Russia (Other)
Responsible Party: Principal Investigator, Diana Vikulova, MD, neurologist, investigator, Clinical Institute of the Brain, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C-fMRI-NBS
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Vegetative State; Stroke; Brain Injury
Keywords: Diagnosed vegetative state after stroke or traumatic brain injury
MeSH Terms: conditions — Persistent Vegetative State; Stroke; Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vegetative state (Experimental): Patients with the diagnosis of the vegetative state
  Interventions: Device: Navigated transcranial magnetic brain stimulation

INTERVENTIONS:
Device: Navigated transcranial magnetic brain stimulation — Standard NBS motor mapping using the Eximia TMS stimulator, Nexstim Ltd., Finland.

SUMMARY:
It has already been demonstrated that mental imagining of the complex motor act, such as limb lifting, can evoke the activation of the involved motor centres even if it doesn't result in movement due to paresis. Aim of the study: using the navigated brain stimulation system create a new diagnostic model for the differential diagnostics between the vegetative state and the minimally conscious state. If the investigators could get from patient the efferent motor response after a verbal command, his level of conscious should not be defined less than the minimally conscious state.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed vegetative state
* age 20-85

Exclusion Criteria:

* oncological history
* cardiac pacemakers and other metal implants
* Modified Ashford Scale scores 3 and more
* predisposing disease with motor neurologic impairment

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
MEP(motor evoked potential) parameter: latency | within the first minute after a verbal command

SECONDARY OUTCOMES:
MEP(motor evoked potential) parameter: amplitude | within the first minute after a verbal command
MEP(motor evoked potential) parameter: motor threshold | within the first minute after a verbal command
conscious state | within the first 6 months after NBS mapping

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Belkin, Prof., MD, Phd, Principal Investigator — Clinical Institute of Brain, Ural State Medical Academy
Locations (1):
- Clinical Institute of Brain, Yekaterinburg, Sverdlovsk Oblast, Russia

REFERENCES:
- See also: Clinical Institute of Brain. Official web-site. — http://www.neuro-ural.ru/
- See also: Nexstim develops, manufactures and markets Navigated Brain Stimulation devices for clinical use and scientific research. — http://www.nexstim.com/